CLINICAL TRIAL: NCT02335957
Title: OPTimizing Irradiation Through Molecular Assessment of Lymph Node (OPTIMAL)
Acronym: OPTIMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo de Investigación Clínica en Oncología Radioterapia (Other)
Responsible Party: Principal Investigator, Esther Prats, ST, Grupo de Investigación Clínica en Oncología Radioterapia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIC-RAD-2014-02
Record Dates: First submitted 2014-12-23; First posted 2015-01-12 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intentional irradiation of lymph nodes (Other): Patients will receive a total dose of 50 Gy in the whole breast and nodal areas(axillary I, II, III, and supraclavicular) with optimization of the technique, in daily fractions of 2 Gy and 5 fractions/week during 5 weeks.
  Interventions: Radiation: Irradiation
- Incidental irradiation of lymph nodes (Experimental): Patients will receive a total dose of 50 Gy in the whole breast, but not aimed at nodal areas, with optimization of the technique, in daily fractions of 2 Gy and 5 fractions/week during 5 weeks.
  Interventions: Radiation: Irradiation

INTERVENTIONS:
Radiation: Irradiation — Intentional versus incidental irradiation of lymphatic node areas, administered using a lineal accelerator, after 3D delimitation of the supraclavicular and axillary levels I, II and III. In both treatment arms, further tumoral bed boost will be allowed according to the investigator criteria, whether dose contribution to the nodal areas can be calculated. Due to its nature, interventions cannot be asked.

SUMMARY:
The main purpose of this study is to show the non-inferiority of the incidental irradiation, as compared to intentional irradiation of the axillary nodes, in terms of 5-years disease-free survival (DFS) of early stage breast cancer patients with limited affectation of sentinel node assessed by OSNA (250 to 15,000 copies/uL), treated with breast-conservative surgery without axillary lymphadenectomy.

DETAILED DESCRIPTION:
Since long, the standard loco-regional treatment of the early-stage breast cancer is breast conservative surgery (tumorectomy) followed by a selective biopsy of the sentinel lymph node and, if positive, lymphadenectomy of axillary levels I and II. Complementary irradiation of the breast and ganglionar areas has shown to reduce disease-specific mortality. Therefore, adjuvant radiotherapy of the whole breast is currently indicated after conservative surgery.

The recommendation to irradiate axillary lymph nodes is clear in patients with more than three affected nodes. The standard volumes to irradiate after lymphadenectomy include supraclavicular and level III axillary regions, while axillary levels I and II, and the internal breast lymph node chain, are reserved for cases of cumbersome axillary affectation, patients who have not undergone lymphadenectomy or it was insufficient, or affectation of the internal breast lymph node chain.

However, when only 1 to 3 nodes are affected, there is no unanimity on the recommendation of radiotherapy, despite some studies have shown that irradiation improves survival. In addition, the National Cancer Institute of Canada trial (NCIC-CTGMA20), high risk patients with negative lymph nodes and patients with positive lymph nodes (most of them with 1 to 3 affected nodes) showed that local irradiation with or without regional lymph node irradiation improved disease-free survival, as well as loco-regional and distant disease control. Moreover, a systematic review including more than 20,000 patients from 45 studies concludes that the irradiation of the breast reduced the loco-regional relapse, even in patients without affected lymph nodes.

One Step Nucleic Acid Amplification (OSNA) is a technique developed by Sysmex Corporation that allows a readily and complete analysis of sentinel lymph nodes during surgery. OSNA provides a quantification of the Cytokeratin 19 (CK19) tumour cell marker in the messenger ribonucleic acid (mRNA) of the sentinel node, the result being expressed as "total tumour load" (TTL), which is a discrete number of copies per microliter. This technique has shown ability to discriminate macrometastasis, micrometastasis or negativity, and to predict affectation of non-sentinel lymph nodes. According to previous results, a TTL < 15,000 is associated with a 85% probability of non-affectation of (non-sentinel) axillar lymph nodes.

The therapeutic value of the axillary lymphadenectomy has been questioned since long, and the recent publication of the Z0011 study proposes solely a selective biopsy of the sentinel lymph node. This has impacted clinical practice guidelines as prestigious as those of the National Comprehensive Cancer Network; however, irradiation is always considered in these cases.

In summary, the amount of nodal volumes to irradiate in early stages of breast cancer is under discussion, particularly in the case of patients not submitted to axillar lymphadenectomy despite affectation of sentinel lymph nodes. In most cases, the irradiation of the breast implies "incidental" irradiation of the axillary level I, and in some cases the level II. For this reason, some groups have decided not to irradiate these axillary regions intentionally, while others advocate irradiating these regions intentionally.

ELIGIBILITY:
Inclusion Criteria:

1. Infiltrating, ductal carcinoma of the breast.
2. Treated with conservative surgery (tumorectomy or quadrantectomy) without lymphadenectomy.
3. Sentinel lymph node assessed by OSNA, with TTL in the range 250 - 15,000 copies/μL.
4. Age ≥ 18 yrs old.
5. Karnofsky Index ≥ 70 %.
6. Signed Informed Consent.

Exclusion Criteria:

1. Other types of breast cancer different from infiltrating ductal carcinoma.
2. Bilateral breast cancer.
3. Males.
4. Mastectomy or axillary homolateral lymph node dissection.
5. Previous thoracic irradiation therapy.
6. Systemic neoadjuvant therapy previous to surgery.
7. Contraindications of radiotherapy (pregnancy, severe collagen diseases).
8. Other neoplasms.
9. Severe associated comorbidities that, according to the investigator criteria, may interfere with the study evaluations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival | 5 years
  The primary outcome will be the 5-years DFS. DFS is defined as the time from randomization to any breast cancer-related event, including local, regional or distant recurrence, or death from breast cancer.

SECONDARY OUTCOMES:
Time to loco-regional recurrence up 5-years | 5 years
  Loco-regional recurrence during the 5-years follow-up, defined as clinical or image-based detection of tumour in treated breast (local recurrence) or in the ipsilateral axilla or supraclavicular fossa (regional recurrence).
Time to distant recurrence up 5-years | 5 years
  Distant recurrence occuring during the 5-years follow-up, defined as defined as clinical or image-based detection of neoplastic affectation of other organs or tissues different from the treated breast, ipsilateral axilla or supraclavicular fossa.
Number of patients with acute toxicity, defined as any adverse event appearing up to one month after finalization of radiotherapy. | 7 years
  Acute toxicity, assessed by a selected subset of the Common Terminology Criteria for Adverse Events v4.0 (CTCAE)
Number of patients with chronic toxicity, defined as any adverse event appearing during follow-up, up to 5 years. | 7 years
  Chronic toxicity , assessed by a selected subset of the Common Terminology Criteria for Adverse Events v4.0 (CTCAE)
Total irradiation dose (Gy) received in axillary levels I, II and III, supraclavicular fossa, and internal mammary chain volumes, at the end of radiotherapy. | 2 years
  Total dose (Gy) received in axillary levels I, II,and II, supraclavicular, and internal mammary chain volumes.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Algara López, Medicine, Principal Investigator — Grupo de Investigación Clínica en Oncología Radioterápica (GICOR)
Locations (50):
- Hospital de Perugia, Perugia, Italy
- Portugal (3):
  - Hospital Espírito Santo, Evora
  - Centro Hospitalar De São João, Porto
  - Hospital Distrital de Santarém, Santarém
- Spain (46):
  - Hospital de Cruces, Barakaldo, Bilbao
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Canary Islands
  - Complejo Hospitalario Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital General Universitario de Santa Lucía, Cartagena, Murcia
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Fundación Hospital de Jove, Gijón, Principality of Asturias
  - Centro Onoclógico de Galicia, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital Universitario de la Ribera, Alzira
  - Hospital Universitario Infanta Cristina, Badajoz
  - Centro Médico Teknon, Barcelona
  - Clínica Platon, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - ICO Duran i Reynals, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Provincial de Castellón, Castelló
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital de Donostia, Donostia / San Sebastian
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de León, León
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Clínico Universitario de San Carlos, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital General Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen de la Macarena, Seville
  - Hospital Virgen del Rocío, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic la Fe, Valencia
  - Instituto Valenciano de Oncología (IVO), Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Hospital Universitario de Araba, Vitoria-Gasteiz
  - Hospital Virgen de la Concha, Zamora
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Background] Kiluk JV, Ly QP, Meade T, Ramos D, Reintgen DS, Dessureault S, Davis M, Shamehdi C, Cox CE. Axillary recurrence rate following negative sentinel node biopsy for invasive breast cancer: long-term follow-up. Ann Surg Oncol. 2011 Dec;18 Suppl 3:S339-42. doi: 10.1245/s10434-009-0704-1. Epub 2009 Sep 24. PMID 19777181
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Darby S, McGale P, Correa C, Taylor C, Arriagada R, Clarke M, Cutter D, Davies C, Ewertz M, Godwin J, Gray R, Pierce L, Whelan T, Wang Y, Peto R. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011 Nov 12;378(9804):1707-16. doi: 10.1016/S0140-6736(11)61629-2. Epub 2011 Oct 19. PMID 22019144
- [Background] Ragaz J, Olivotto IA, Spinelli JJ, Phillips N, Jackson SM, Wilson KS, Knowling MA, Coppin CM, Weir L, Gelmon K, Le N, Durand R, Coldman AJ, Manji M. Locoregional radiation therapy in patients with high-risk breast cancer receiving adjuvant chemotherapy: 20-year results of the British Columbia randomized trial. J Natl Cancer Inst. 2005 Jan 19;97(2):116-26. doi: 10.1093/jnci/djh297. PMID 15657341
- [Background] Overgaard M, Nielsen HM, Overgaard J. Is the benefit of postmastectomy irradiation limited to patients with four or more positive nodes, as recommended in international consensus reports? A subgroup analysis of the DBCG 82 b&c randomized trials. Radiother Oncol. 2007 Mar;82(3):247-53. doi: 10.1016/j.radonc.2007.02.001. Epub 2007 Feb 15. PMID 17306393
- [Background] van Wely BJ, Teerenstra S, Schinagl DA, Aufenacker TJ, de Wilt JH, Strobbe LJ. Systematic review of the effect of external beam radiation therapy to the breast on axillary recurrence after negative sentinel lymph node biopsy. Br J Surg. 2011 Mar;98(3):326-33. doi: 10.1002/bjs.7360. Epub 2010 Nov 30. PMID 21254004
- [Background] Peg V, Espinosa-Bravo M, Vieites B, Vilardell F, Antunez JR, de Salas MS, Delgado-Sanchez JJ, Pinto W, Gozalbo F, Petit A, Sansano I, Del Mar Tellez M, Rubio IT. Intraoperative molecular analysis of total tumor load in sentinel lymph node: a new predictor of axillary status in early breast cancer patients. Breast Cancer Res Treat. 2013 May;139(1):87-93. doi: 10.1007/s10549-013-2524-z. Epub 2013 Apr 11. PMID 23576079
- [Background] Veronesi U, Orecchia R, Zurrida S, Galimberti V, Luini A, Veronesi P, Gatti G, D'Aiuto G, Cataliotti L, Paolucci R, Piccolo P, Massaioli N, Sismondi P, Rulli A, Lo Sardo F, Recalcati A, Terribile D, Acerbi A, Rotmensz N, Maisonneuve P. Avoiding axillary dissection in breast cancer surgery: a randomized trial to assess the role of axillary radiotherapy. Ann Oncol. 2005 Mar;16(3):383-8. doi: 10.1093/annonc/mdi089. Epub 2005 Jan 24. PMID 15668261
- [Background] Martelli G, Boracchi P, De Palo M, Pilotti S, Oriana S, Zucali R, Daidone MG, De Palo G. A randomized trial comparing axillary dissection to no axillary dissection in older patients with T1N0 breast cancer: results after 5 years of follow-up. Ann Surg. 2005 Jul;242(1):1-6; discussion 7-9. doi: 10.1097/01.sla.0000167759.15670.14. PMID 15973094
- [Background] Hwang RF, Gonzalez-Angulo AM, Yi M, Buchholz TA, Meric-Bernstam F, Kuerer HM, Babiera GV, Tereffe W, Liu DD, Hunt KK. Low locoregional failure rates in selected breast cancer patients with tumor-positive sentinel lymph nodes who do not undergo completion axillary dissection. Cancer. 2007 Aug 15;110(4):723-30. doi: 10.1002/cncr.22847. PMID 17587208
- [Background] Bilimoria KY, Bentrem DJ, Hansen NM, Bethke KP, Rademaker AW, Ko CY, Winchester DP, Winchester DJ. Comparison of sentinel lymph node biopsy alone and completion axillary lymph node dissection for node-positive breast cancer. J Clin Oncol. 2009 Jun 20;27(18):2946-53. doi: 10.1200/JCO.2008.19.5750. Epub 2009 Apr 13. PMID 19364968
- [Background] Veronesi U, Viale G, Paganelli G, Zurrida S, Luini A, Galimberti V, Veronesi P, Intra M, Maisonneuve P, Zucca F, Gatti G, Mazzarol G, De Cicco C, Vezzoli D. Sentinel lymph node biopsy in breast cancer: ten-year results of a randomized controlled study. Ann Surg. 2010 Apr;251(4):595-600. doi: 10.1097/SLA.0b013e3181c0e92a. PMID 20195151
- [Background] Caudle AS, Hunt KK, Kuerer HM, Meric-Bernstam F, Lucci A, Bedrosian I, Babiera GV, Hwang RF, Ross MI, Feig BW, Hoffman K, Litton JK, Sahin AA, Yang W, Hortobagyi GN, Buchholz TA, Mittendorf EA. Multidisciplinary considerations in the implementation of the findings from the American College of Surgeons Oncology Group (ACOSOG) Z0011 study: a practice-changing trial. Ann Surg Oncol. 2011 Sep;18(9):2407-12. doi: 10.1245/s10434-011-1593-7. No abstract available. PMID 21327455
- [Background] Giuliano AE, McCall L, Beitsch P, Whitworth PW, Blumencranz P, Leitch AM, Saha S, Hunt KK, Morrow M, Ballman K. Locoregional recurrence after sentinel lymph node dissection with or without axillary dissection in patients with sentinel lymph node metastases: the American College of Surgeons Oncology Group Z0011 randomized trial. Ann Surg. 2010 Sep;252(3):426-32; discussion 432-3. doi: 10.1097/SLA.0b013e3181f08f32. PMID 20739842
- [Background] Giuliano AE, Hunt KK, Ballman KV, Beitsch PD, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, McCall LM, Morrow M. Axillary dissection vs no axillary dissection in women with invasive breast cancer and sentinel node metastasis: a randomized clinical trial. JAMA. 2011 Feb 9;305(6):569-75. doi: 10.1001/jama.2011.90. PMID 21304082
- [Background] Carlson RW, Hudis CA, Pritchard KI; National Comprehensive Cancer Network Breast Cancer Clinical Practice Guidelines in Oncology; American Society of Clinical Oncology Technology Assessment on the Use of Aromatase Inhibitors; St Gallen International Expert Consensus on the Primary Therapy of Early Breast Cancer. Adjuvant endocrine therapy in hormone receptor-positive postmenopausal breast cancer: evolution of NCCN, ASCO, and St Gallen recommendations. J Natl Compr Canc Netw. 2006 Nov;4(10):971-9. doi: 10.6004/jnccn.2006.0082. PMID 17112447
- [Background] Setton J, Cody H, Tan L, Morrow M, Hudis C, Catalano J, McCormick B, Powell S, Ho A. Radiation field design and regional control in sentinel lymph node-positive breast cancer patients with omission of axillary dissection. Cancer. 2012 Apr 15;118(8):1994-2003. doi: 10.1002/cncr.26504. Epub 2011 Aug 31. PMID 21882186
- [Background] Haffty BG, Hunt KK, Harris JR, Buchholz TA. Positive sentinel nodes without axillary dissection: implications for the radiation oncologist. J Clin Oncol. 2011 Dec 1;29(34):4479-81. doi: 10.1200/JCO.2011.36.1667. Epub 2011 Oct 31. No abstract available. PMID 22042942
- [Background] Bayo E, Herruzo I, Arenas M, Algara M. Consensus on the regional lymph nodes irradiation in breast cancer. Clin Transl Oncol. 2013 Oct;15(10):766-73. doi: 10.1007/s12094-013-1027-z. Epub 2013 Mar 22. PMID 23519538
- [Derived] Algara M, Rodriguez E, Martinez-Arcelus FJ, Salinas J, Sanz X, Beato I, Manso A, Soler A, Rodriguez JR, Frias A, Calin A, Juan G, Meireles P, Flaquer A; OPTIMAL investigators. OPTimizing Irradiation through Molecular Assessment of Lymph node (OPTIMAL): a randomized clinical trial. Radiother Oncol. 2022 Nov;176:76-82. doi: 10.1016/j.radonc.2022.09.006. Epub 2022 Sep 19. PMID 36210628
- [Derived] Algara Lopez M, Rodriguez Garcia E, Beato Tortajada I, Martinez Arcelus FJ, Salinas Ramos J, Rodriguez Garrido JR, Sanz Latiesas X, Soler Rodriguez A, Juan Rijo G, Flaquer Garcia A. OPTimizing Irradiation through Molecular Assessment of Lymph node (OPTIMAL): a randomized open label trial. Radiat Oncol. 2020 Oct 2;15(1):229. doi: 10.1186/s13014-020-01672-7. PMID 33008422